CLINICAL TRIAL: NCT02486003
Title: The Use of a Portable 3D Head Mounted Display (HMD) With Integrated Eye Capture Technology for the Diagnosis of Dizziness Associated With Mild Traumatic Brain Injury (mTBI)
Brief Title: Testing mTBI in Athletes
Status: Completed | Type: Observational
Sponsor: University of Miami (Other)
Collaborators: National Football League (Other)
Responsible Party: Principal Investigator, Michael E. Hoffer, Professor of Otolaryngology, University of Miami
Other Study IDs: 20150361
Record Dates: First submitted 2015-06-26; First posted 2015-06-30 (Estimated); Last update posted 2017-12-22 (Actual); Status verified 2017-12

CONDITIONS: Mild Traumatic Brain Injury; Brain Concussion
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- mTBI athletes: College athletes who undergo an mTBI during the season
- Control athletes: College athletes who do not undergo an mTBI during the season
- Control non-athletes: Control non-athletes with long term follow-up of approximately 4-6 weeks and 3-5 months

SUMMARY:
This study will assess the effectiveness of a portable goggle system in the diagnosis of mild traumatic brain injury (mTBI) in athletes.

DETAILED DESCRIPTION:
The purpose of this research study is to assess oculomotor, vestibular and reaction time responses in mild traumatic brain injury (mTBI) athletes, as well as healthy individuals. These measurements will be recorded using a portable goggle system (IPAS). The goal is to determine whether this IPAS goggle system is effective at diagnosing mTBI. A secondary goal is to determine whether this IPAS goggle system is effective at ruling out the diagnosis of mTBI in athletes and non-athletes that do not have the condition.

The IPAS is a portable 3D head mounted display. The IPAS goggles are programmed with a series of tests that track eye motions in response to a target. This device has been determined to be a Non-Significant Risk to study participants.

There are three groups of interest in this study: athletes who suffer an mTBI, athletes who do have an mTBI, and healthy non-athletes.

ELIGIBILITY:
Inclusion Criteria:

* Males and females from 18 - 40 years of age who participate in intercollegiate athletics at the University of Miami to include all levels of sports whether NCAA or club. Initial recruitment will include high intensity sports alone (these include but are not limited to football, Men's and Women's Soccer, Men's and Women's Basketball, Men's Baseball and Women's Softball, and club sports to include Men's and Women's Lacrosse, Hockey, Rugby, and Field Hockey).

Exclusion Criteria:

* History of brain injury resulting from a penetrating wound to the head.
* Presence of severe aphasia
* History of diagnosed neuropsychiatric disorders (e.g. hypochondriasis, major depression, schizophrenia
* Documented neurodegenerative disorders
* Pregnancy, [Female candidates will be asked if they are pregnant]
* Prior disorders of hearing and balance including:

  1. Meniere's disease
  2. Multiple sclerosis
  3. Vestibular neuritis
  4. Vestibular schwannoma
  5. Sudden sensorineural hearing loss
* Cerebrovascular disorders
* History of ear operation other than myringotomy tube in the past
* Systemic disorders: e.g. chronic renal failure, cirrhosis of the liver, etc.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects will be recruited from the population of athletes in the intercollege athletic programs at the University of Miami. This will include athletes in NCAA Sports as well as intercollege club sports. Aged and sex matched controls will be collected from the general student body of the University of Miami.
Sampling Method: Non-Probability Sample
Enrollment: 329 (Actual)
Dates: Start 2015-05; Primary Completion 2017-08-14 (Actual); Study Completion 2017-08-14 (Actual)

PRIMARY OUTCOMES:
Vestibular, oculomotor, and reaction time test results | 3 months
  IPAS testing will be conducted by placing the IPAS goggles on the head of a patient and asking the patient to follow instructions while a set of tests is performed. Each of these tests simply involves eye motions in response to a target.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Miami Miller School of Medicine, Miami, Florida, United States